CLINICAL TRIAL: NCT05261009
Title: PENG Block Versus LP Block for Postoperative Analgesia After Anterior Total Hip
Brief Title: PENG Block Versus LP Block for THA Postop Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00078699
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Hip Pain Chronic
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peri-capsular Nerve Group (PENG) (Experimental): Those subjects assigned to the PENG treatment arm will receive a PENG block using 20mL of 0.2% ropivacaine with 1:400,000 epinephrine dosed in 5mL increments with negative aspiration beforehand and between each aliquot.
  Interventions: Drug: Peri-capsular Nerve Group (PENG)
- Lumbar Plexus Block (LPB) (Active Comparator): Those subjects assigned to the LPB treatment arm will receive a stimulation-based LPB dosed with 20cc of 0.2% ropivacaine with 1:400,000 dilution epinephrine dosed in 5mL increments with negative aspiration beforehand and between each aliquot.
  Interventions: Other: Lumbar Plexus Block (LPB)

INTERVENTIONS:
Drug: Peri-capsular Nerve Group (PENG) — PENG block for postoperative pain management
  Arms: Peri-capsular Nerve Group (PENG)
Other: Lumbar Plexus Block (LPB) — LPB for postoperative pain management
  Arms: Lumbar Plexus Block (LPB)

SUMMARY:
The purpose of this randomized, double blinded, prospective study is to compare the postoperative analgesia provided by the PENG block to that provided by the LPB for patients undergoing primary anterior approach THA.

DETAILED DESCRIPTION:
Regional anesthesia procedures represent a common modality for postoperative analgesia after total hip arthroplasty surgeries (THA). The standard practice many years has been the Lumbar Plexus block (LPB), which anesthetizes the L1-L5 lumbar nerve roots1. While the LPB offers analgesia from the associated sensory block, it also blocks motor fibers, leading to lower extremity weakness that could potentially delay the patient's ability to participate in early physical therapy and may thereby delay discharge. In the past several years, newer regional anesthesia block approaches have been described and investigated in an attempt to provide patients with postoperative analgesia while avoiding associated muscle weakness, facilitating earlier physical therapy participation and discharge. One such nerve block is the peri-capsular nerve group (PENG) block, which anesthetizes the articular branches of the femoral, obturator, and accessory obturator nerves providing sensory innervation to the hip joint capsule without consistently causing lower extremity weakness2. Some institutions are utilizing the PENG block to provide postoperative analgesia and facilitate early mobilization. There are currently no prospective studies that directly compare the efficacy of LPB to PENG block for providing postoperative analgesia after THA.

ELIGIBILITY:
Inclusion Criteria:

* elective primary total hip arthroplasty surgery anterior approach
* provided informed consent
* no contraindications to medications used in providing the analgesic blocks

Exclusion Criteria:

* contraindications to regional anesthesia, such as an allergy to amide local anesthetics
* pre-existing coagulopathy or thrombocytopenia <100,000
* refusal of analgesic block for pain management
* presence of an progressive lower extremity neurological deficit
* localized or systemic infection
* chronic use of high dose opioid analgesics (defined as daily use greater than 60 mg oxycodone equivalents)
* pregnant
* refusal of consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rawad Hamzi, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Started | 76 | 76
Completed | 75 | 75
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB) | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 62
  >=65 years | 46 | 44 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 43 | 91
  Male | 28 | 33 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 74 | 73 | 147
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 69 | 71 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 76 | 76 | 152

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Pain Score
Description: a comparison of patient-reported numeric rating scale (NRS) pain scores with movement at six hours following block placement. Equivalency will be defined as a difference of less than one point in either direction on the eleven-point NRS pain scale. Score ranges from 0-10 with a higher score denoting more pain.
Time Frame: hour 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 75 | 75
units on a scale | 4.0 (2.8) | 2.8 (2.4)

2. Secondary Outcome: NRS Pain Score
Description: a comparison of patient-reported numeric rating scale (NRS) pain scores with movement at 12 hours following block placement. Score ranges from 0-10 with a higher score denoting more pain.
Time Frame: hour 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 75 | 75
units on a scale | 6.1 (2.4) | 5.0 (2.5)

3. Secondary Outcome: NRS Pain Score
Description: a comparison of patient-reported numeric rating scale (NRS) pain scores with movement at 18 hours following block placement. Score ranges from 0-10 with a higher score denoting more pain.
Time Frame: hour 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 75 | 75
units on a scale | 6.0 (2.8) | 5.3 (2.5)

4. Secondary Outcome: NRS Pain Score
Description: a comparison of patient-reported numeric rating scale (NRS) pain scores with movement at 24 hours following block placement. Score ranges from 0-10 with a higher score denoting more pain.
Time Frame: hour 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 75 | 75
units on a scale | 5.7 (2.2) | 4.6 (2.2)

5. Secondary Outcome: Time in Minutes Until Opioid Administration
Description: Time to first dose of opioid rescue for postoperative pain management - This outcome was evaluated in time to first opioid dose, which was measured in hours - no analysis for mean, median, or any of the others suggested - It was calculated as time of block to time of first opioid dose-hours and minutes.
Time Frame: hour 24
Population: The number analyzed for pain meds in each group is different from the participant flow because not everyone had to have opioids within the first 24 hours. This outcome is related to only those that required opioids in each group.
Measure: Mean (Standard Deviation); unit: minutes until first dose
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 72 | 70
minutes until first dose | 464.98 (221.67) | 394.69 (158.39)

6. Secondary Outcome: Motor Strength
Description: straight leg raise at 6 hours after block placed rated on a 0-5 scale with a higher score indicating better movement
Time Frame: hour 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 75 | 75
units on a scale | 3.5 (1.6) | 2.4 (1.3)

7. Secondary Outcome: Distance Ambulated
Description: Recorded in feet during first physical therapy
Time Frame: hour 24
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 75 | 75
feet | 59.1 (49.6) | 43.9 (42.2)

ADVERSE EVENTS:
Time Frame: 24 hour follow up of evaluating adverse events
Arm/Group | Peri-capsular Nerve Group (PENG) | Lumbar Plexus Block (LPB)
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/75 | 2/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peri-capsular Nerve Group (PENG) (N=75) | Lumbar Plexus Block (LPB) (N=75)
Right hip dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pumonary embolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
epidural spread (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — LP block inadvertently spread into the epidural space

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT05261009/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT05261009/ICF_002.pdf